CLINICAL TRIAL: NCT06935240
Title: Investigation of Effects of External Electrical Stimulation in Women With Vaginal Laxity
Brief Title: Investigation of Effects of Electrical Stimulation in Women With Vaginal Laxity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other); Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zehra KORKUT, Assistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/190
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Individuals who meet the inclusion criteria and sign the consent form will be randomly divided into 3 groups (Control, Neuromuscular ES, TENS). Randomization will be performed by a researcher who is not involved in the study using computer-assisted randomization blocks.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients in this group will receive only lifestyle recommendations (fluid consumption, diet, weight gain, constipation and bladder irritations) to maintain urinary control.
- Nöromusculer Es (Experimental): The neuromuscular ES wearable device INNOVO® (Atlantic Therapeutics, Galway, Ireland) will be used three days a week in the supine hook position with urge mode (program 2: 10 Hz frequency, 250 ms pulse width, 0.5 seconds acceleration and deceleration times, 5 seconds contraction time and 0 seconds parameters) along with lifestyle recommendations. The device will be glued around the hip/pelvis of the patients so that the electrodes will coincide with the anterior and posterior of the right and left hip, the right-left pelvic side and the right-left gluteal region. The application will take 30 minutes.
  Interventions: Device: Treatment
- Tens (Experimental): A current with a pulse width of 200 milliseconds and a frequency of 10 Hz will be applied three days a week in the prone position with a parasacral TENS device (Intelect, economy) along with lifestyle recommendations. Electrodes will be placed bilaterally and parasacrally. The application will last 30 minutes.
  Interventions: Device: Treatment

INTERVENTIONS:
Device: Treatment — Nöromusculer and Transcutaneus Electrical Neuron stimulations
  Arms: Nöromusculer Es; Tens

SUMMARY:
The purpose of this study is to compare the effects of different externally applied electrical stimulation methods on overactive bladder (OAB) symptoms, quality of life, and patients' perception of improvement.

DETAILED DESCRIPTION:
Current treatment options in the management of AAM are graded into 4 steps by various clinical guidelines. The first step consists of behavioral treatment methods such as lifestyle modification and bladder training and physiotherapy and rehabilitation approaches. Physiotherapy and rehabilitation approaches include various techniques such as pelvic floor muscle training, electrical stimulation (ES), manual therapy and kinesio taping. Transcutaneous electrical nerve stimulation (TENS) is a non-invasive therapeutic method commonly preferred for acute and chronic pain management.

The purpose of TENS in the management of AAM is one of the external ES methods used to inhibit presynaptic afferent neurons carrying impulses from the bladder by stimulating peripheral segmental dermatome nerves. Thus, TENS can affect neural pathways that modulate afferent/efferent impulses in the spinal and supraspinal areas. The portable TENS device is a two-channel output device with self-adhesive electrodes and adjustable treatment frequency and duration. The device is used in AAM by selecting 200 millisecond pulse width and 10 hz frequency parameters. With this frequency, related neural pathways can be modulated and detrusor overactivity can be controlled.

Neuromuscular ES (Innovo ®) (Atlantic Therapeutics, Galway, Ireland), which can be used as external ES in the treatment of AAM, is a new neuromuscular ES device developed to retrain the pelvic floor muscles and inhibit the detrusor muscle through electrodes placed in a garment in the treatment of incontinence. In the literature, this device is also known as a type of external ES application (new generation external ES) applied over the pelvis/hip and can be easily worn and used by the patient. This device is attached to a 2-piece wrapped garment that holds the four electrodes in place in the pelvis/hip with hydrogel adhesive. Program 2 was designed in this device for the presence of urge/pinch type incontinence. This program includes 10 Hz frequency, 250 ms pulse width, 0.5 seconds acceleration and deceleration times, 5 seconds contraction time and 0 seconds parameters. With this program, the nerve controlling the pelvic floor muscle mechanism is stimulated and detrusor overactivity can be controlled.

While tibial nerve stimulation has been mostly used in patients with AAM, it has recently been observed that external ES applications have started to be applied alone or in combination with other treatments. When the literature is reviewed, it is seen that there are a limited number of external ES applications in patients with AAM, but there is no study comparing these applications. Therefore, the aim of this study was to compare the effects of different external ES applications on bladder functions, AAM symptoms, quality of life and patients' perception of recovery in women with AAM. In this sense, it is thought that our study will contribute to the literature and will have original value.

ELIGIBILITY:
Inclusion Criteria:

To be between the ages of 18-65 Being diagnosed with AAM Volunteer Becoming literate

Exclusion Criteria:

Sensory loss Presence of infection Having a pacemaker Metal implant presence Malignancy story Having serious cardiovascular problems Presence of severe pelvic organ prolapse (above stage 2) Pregnancy presence Lumbosacral peripheral nerve lesion

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Symptom severity Overactive Bladder-V8 Questionnaire (OAB-V8) | 6 weeks

SECONDARY OUTCOMES:
bladder diary results | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)